CLINICAL TRIAL: NCT03814824
Title: Volumetric Laser Endomicroscopy With Intelligent Real-time Image Segmentation (IRIS): a Multi-center Randomized Prospective Study
Brief Title: Volumetric Laser Endomicroscopy With Intelligent Real-time Image Segmentation (IRIS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: NinePoint Medical (Industry); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-0963
Record Dates: First submitted 2019-01-08; First posted 2019-01-24 (Actual); Results first posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-09

CONDITIONS: Barrett's Esophagus Without Dysplasia; Barrett's Esophagus With Dysplasia; Barrett's Esophagus With Low Grade Dysplasia; Barrett's Esophagus With High Grade Dysplasia; Barrett's Esophagus With Dysplasia, Unspecified
Keywords: VLE; Volumetric laser endomicroscopy; IRIS; Intelligent real-time image segmentation; Barrett's Esophagus
MeSH Terms: conditions — Barrett Esophagus | interventions — Genes, BRCA1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- VLE without IRIS, followed by VLE with IRIS (Active Comparator): VLE (Volumetric laser endomicroscopy) performed alone, followed by IRIS (Intelligent real-time image segmentation) imaging.
  Interventions: Diagnostic Test: IRIS (Intelligent real-time image segmentation); Diagnostic Test: VLE (Volumetric laser endomicroscopy)
- VLE with IRIS, followed by VLE without IRIS (Active Comparator): VLE (Volumetric laser endomicroscopy) performed with IRIS (Intelligent real-time image segmentation) imaging, followed by VLE alone.
  Interventions: Diagnostic Test: IRIS (Intelligent real-time image segmentation); Diagnostic Test: VLE (Volumetric laser endomicroscopy)

INTERVENTIONS:
Diagnostic Test: IRIS (Intelligent real-time image segmentation) — IRIS has the ability to identify and display three specific images features that may correlate with dysplasia that are represented in different color schemes.
Diagnostic Test: VLE (Volumetric laser endomicroscopy) — VLE uses infrared light to produce real time high-resolution cross sectional imaging of the esophagus.

SUMMARY:
This is a prospective randomized clinical trial examining how IRIS (Intelligent Real-time Image Segmentation) affects biopsy patterns in VLE (Volumetric laser endomicroscopy).

DETAILED DESCRIPTION:
Patients will undergo a VLE exam with and without IRIS per the standard of care. All patients regardless of the study participation in this study would receive VLE with and without IRIS clinically. They will be randomized into VLE without IRIS first vs VLE with IRIS first. The BUDDY Randomization System, provided for use by the Northwell Health Biostatistics Unit, will be used for this. Randomization will be stratified based on prior diagnosis of dysplasia. The order in which the patient is randomized to will be recorded on the case report form. There will be concealed allocation as the study coordinator performing the randomization will not know the order of the next allocation.

Both VLE and IRIS imaging are being performed as standard of care. However, randomization of the order allows for comparison of the two. Regions of interest (ROI) will be recorded using a full scan and recorded on the case report form. The time to identification of ROIs will also be recorded. Each group will then cross over such that the VLE without IRIS group will then have IRIS turned on. ROI will then be recorded for each group based on full scans. A consensus ROI will be recorded based on the two exams. Only one ROI per centimeter will be allowed to avoid overlapping of laser marks. In addition, VLE without IRIS and IRIS marks within 75 frames of each other or 2 hours (on a clock face orientation) will be considered the same target.

Laser marking will then be performed. A double laser mark will be applied to all IRIS ROIs. A single laser mark will be applied to VLE ROIs. Targeted biopsies will be taken of all laser marks and placed in separate biopsy jars. Biopsies will be taken in between the laser marks for double laser marked areas. For single laser marks, biopsies will be taken on either side of the laser mark. Resection of visible lesions will then occur per standard of care (if present) followed by random biopsies of the segment. Random biopsies are pinch biopsies every 1 cm the length of the Barrett's in a 4 quadrant fashion per gastrointestinal society guidelines. There are no additional research biopsies being performed outside this study. The targeted biopsies are based on the VLE features that are suspicious for dysplasia and thus standard of care. The other biopsies being performed here are random biopsies which are also being performed for standard of care. Biopsied samples will be stored per standard of care procedures per the pathology department. They will not be stored for future research purposes.

Following each procedure, the physician will be asked a series of Likert Scale questions to assess the utility of IRIS in that procedure, including how it impacts their confidence in image interpretation, their ability to assimilate data more easily and quickly, and their overall perception of the technology.

Although, the VLE with IRIS and VLE without IRIS are being performed as standard of care, all adverse events will be recorded and reported to the IRB.

All data will be entered into a central encrypted REDCap database.

Expert pathologists who specialize in gastrointestinal pathology will read the histology. A second gastrointestinal pathologist will confirm any histologic diagnosis of dysplasia. This is the standard of care at Northwell Health and academic medical centers per gastrointestinal society guidelines.

All procedures (upper endoscopy, volumetric laser endomicroscopy, and IRIS enhanced VLE) will be performed as standard of care. The prospective data collection and initial randomization will be the research component. All data collected will be de-identified before being transferred into a database. This will be kept in a safe place that is only accessible to the research team.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at the time of informed consent
* Barrett's esophagus greater than 2 cm in length
* Undergoing a scheduled upper endoscopy with VLE exam for surveillance as standard of care

Exclusion Criteria:

* Less than 18 years old at the time of informed consent
* Unable to provide written informed consent
* Esophageal stenosis/stricture preventing VLE
* Esophagitis
* Severe medical comorbidities preventing endoscopy
* Pregnancy
* Uncontrolled coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2021-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arvind Trindade, MD, Principal Investigator — Northwell Health
Locations (3):
- United States (3):
  - Mayo Clinic, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota
  - North Shore University Hospital, Manhasset, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shaheen NJ, Falk GW, Iyer PG, Gerson LB; American College of Gastroenterology. ACG Clinical Guideline: Diagnosis and Management of Barrett's Esophagus. Am J Gastroenterol. 2016 Jan;111(1):30-50; quiz 51. doi: 10.1038/ajg.2015.322. Epub 2015 Nov 3. PMID 26526079
- [Background] Spechler SJ, Souza RF. Barrett's esophagus. N Engl J Med. 2014 Aug 28;371(9):836-45. doi: 10.1056/NEJMra1314704. No abstract available. PMID 25162890
- [Background] Pohl H, Welch HG. The role of overdiagnosis and reclassification in the marked increase of esophageal adenocarcinoma incidence. J Natl Cancer Inst. 2005 Jan 19;97(2):142-6. doi: 10.1093/jnci/dji024. PMID 15657344
- [Background] Bhat SK, McManus DT, Coleman HG, Johnston BT, Cardwell CR, McMenamin U, Bannon F, Hicks B, Kennedy G, Gavin AT, Murray LJ. Oesophageal adenocarcinoma and prior diagnosis of Barrett's oesophagus: a population-based study. Gut. 2015 Jan;64(1):20-5. doi: 10.1136/gutjnl-2013-305506. Epub 2014 Apr 3. PMID 24700439
- [Background] Corley DA, Mehtani K, Quesenberry C, Zhao W, de Boer J, Weiss NS. Impact of endoscopic surveillance on mortality from Barrett's esophagus-associated esophageal adenocarcinomas. Gastroenterology. 2013 Aug;145(2):312-9.e1. doi: 10.1053/j.gastro.2013.05.004. Epub 2013 May 11. PMID 23673354
- [Background] Levine DS, Haggitt RC, Blount PL, Rabinovitch PS, Rusch VW, Reid BJ. An endoscopic biopsy protocol can differentiate high-grade dysplasia from early adenocarcinoma in Barrett's esophagus. Gastroenterology. 1993 Jul;105(1):40-50. doi: 10.1016/0016-5085(93)90008-z. PMID 8514061
- [Background] Jankowski M, Wani S. Diagnostic and Management Implications of Basic Science Advances in Barrett's Esophagus. Curr Treat Options Gastroenterol. 2015 Mar;13(1):16-29. doi: 10.1007/s11938-014-0040-9. PMID 25567106
- [Background] Trindade AJ, Smith MS, Pleskow DK. The new kid on the block for advanced imaging in Barrett's esophagus: a review of volumetric laser endomicroscopy. Therap Adv Gastroenterol. 2016 May;9(3):408-16. doi: 10.1177/1756283X16639003. Epub 2016 Mar 21. PMID 27134668
- [Background] Wolfsen HC, Sharma P, Wallace MB, Leggett C, Tearney G, Wang KK. Safety and feasibility of volumetric laser endomicroscopy in patients with Barrett's esophagus (with videos). Gastrointest Endosc. 2015 Oct;82(4):631-40. doi: 10.1016/j.gie.2015.03.1968. Epub 2015 May 6. PMID 25956472
- [Background] Trindade AJ, Leggett CL, Chang KJ. Volumetric laser endomicroscopy in the management of Barrett's esophagus. Curr Opin Gastroenterol. 2017 Jul;33(4):254-260. doi: 10.1097/MOG.0000000000000366. PMID 28402993
- [Background] Swager AF, de Groof AJ, Meijer SL, Weusten BL, Curvers WL, Bergman JJ. Feasibility of laser marking in Barrett's esophagus with volumetric laser endomicroscopy: first-in-man pilot study. Gastrointest Endosc. 2017 Sep;86(3):464-472. doi: 10.1016/j.gie.2017.01.030. Epub 2017 Feb 2. PMID 28161451
- [Background] Swager AF, Tearney GJ, Leggett CL, van Oijen MGH, Meijer SL, Weusten BL, Curvers WL, Bergman JJGHM. Identification of volumetric laser endomicroscopy features predictive for early neoplasia in Barrett's esophagus using high-quality histological correlation. Gastrointest Endosc. 2017 May;85(5):918-926.e7. doi: 10.1016/j.gie.2016.09.012. Epub 2016 Sep 19. PMID 27658906
- [Background] Leggett CL, Gorospe EC, Chan DK, Muppa P, Owens V, Smyrk TC, Anderson M, Lutzke LS, Tearney G, Wang KK. Comparative diagnostic performance of volumetric laser endomicroscopy and confocal laser endomicroscopy in the detection of dysplasia associated with Barrett's esophagus. Gastrointest Endosc. 2016 May;83(5):880-888.e2. doi: 10.1016/j.gie.2015.08.050. Epub 2015 Sep 3. PMID 26344884
- [Background] Trindade AJ, Vamadevan AS, Sejpal DV. Finding a needle in a haystack: use of volumetric laser endomicroscopy in targeting focal dysplasia in long-segment Barrett's esophagus. Gastrointest Endosc. 2015 Oct;82(4):756; discussion 757. doi: 10.1016/j.gie.2015.03.1984. Epub 2015 May 21. No abstract available. PMID 26005011
- [Background] Trindade AJ, George BJ, Berkowitz J, Sejpal DV, McKinley MJ. Volumetric laser endomicroscopy can target neoplasia not detected by conventional endoscopic measures in long segment Barrett's esophagus. Endosc Int Open. 2016 Mar;4(3):E318-22. doi: 10.1055/s-0042-101409. PMID 27004250
- [Background] Leggett CL, Gorospe E, Owens VL, Anderson M, Lutzke L, Wang KK. Volumetric laser endomicroscopy detects subsquamous Barrett's adenocarcinoma. Am J Gastroenterol. 2014 Feb;109(2):298-9. doi: 10.1038/ajg.2013.422. No abstract available. PMID 24496431
- [Background] Swager AF, Boerwinkel DF, de Bruin DM, Faber DJ, van Leeuwen TG, Weusten BL, Meijer SL, Bergman JJ, Curvers WL. Detection of buried Barrett's glands after radiofrequency ablation with volumetric laser endomicroscopy. Gastrointest Endosc. 2016 Jan;83(1):80-8. doi: 10.1016/j.gie.2015.05.028. Epub 2015 Jun 26. PMID 26124075
- [Background] Trindade AJ, Sideridis K, Thomas RM. Buried Barrett's Esophagus Presenting as a Subepithelial Nodule. Am J Gastroenterol. 2016 Oct;111(10):1378. doi: 10.1038/ajg.2016.242. No abstract available. PMID 27694877
- [Background] Mashimo H. Subsquamous intestinal metaplasia after ablation of Barrett's esophagus: frequency and importance. Curr Opin Gastroenterol. 2013 Jul;29(4):454-9. doi: 10.1097/MOG.0b013e3283622796. PMID 23674187
- [Background] Atkinson C, Singh S, Fisichella PM. Volumetric laser endomicroscopy in the detection of neoplastic lesions of the esophagus. Dig Liver Dis. 2016 Jun;48(6):692. doi: 10.1016/j.dld.2016.02.013. Epub 2016 Mar 2. No abstract available. PMID 26976783
- [Background] Alshelleh M, Inamdar S, McKinley M, Stewart M, Novak JS, Greenberg RE, Sultan K, Devito B, Cheung M, Cerulli MA, Miller LS, Sejpal DV, Vegesna AK, Trindade AJ. Incremental yield of dysplasia detection in Barrett's esophagus using volumetric laser endomicroscopy with and without laser marking compared with a standardized random biopsy protocol. Gastrointest Endosc. 2018 Jul;88(1):35-42. doi: 10.1016/j.gie.2018.01.032. Epub 2018 Feb 2. PMID 29410080
- [Background] Trindade AJ, Inamdar S, Smith MS, Chang KJ, Leggett CL, Lightdale CJ, Pleskow DK, Sejpal DV, Tearney GJ, Thomas RM, Wallace MB. Volumetric laser endomicroscopy in Barrett's esophagus: interobserver agreement for interpretation of Barrett's esophagus and associated neoplasia among high-frequency users. Gastrointest Endosc. 2017 Jul;86(1):133-139. doi: 10.1016/j.gie.2016.11.026. Epub 2016 Nov 27. PMID 27899321
- [Background] Trindade AJ, Inamdar S, Smith MS, Rosen L, Han D, Chang KJ, Leggett CL, Lightdale CJ, Pleskow DK, Sejpal DV, Tearney GJ, Thomas RM, Wallace MB. Learning curve and competence for volumetric laser endomicroscopy in Barrett's esophagus using cumulative sum analysis. Endoscopy. 2018 May;50(5):471-478. doi: 10.1055/s-0043-121569. Epub 2017 Nov 27. PMID 29179229
- [Background] Evans JA, Poneros JM, Bouma BE, Bressner J, Halpern EF, Shishkov M, Lauwers GY, Mino-Kenudson M, Nishioka NS, Tearney GJ. Optical coherence tomography to identify intramucosal carcinoma and high-grade dysplasia in Barrett's esophagus. Clin Gastroenterol Hepatol. 2006 Jan;4(1):38-43. doi: 10.1053/S1542-3565(05)00746-9. PMID 16431303
- [Background] Swager AF, van der Sommen F, Klomp SR, Zinger S, Meijer SL, Schoon EJ, Bergman JJGHM, de With PH, Curvers WL. Computer-aided detection of early Barrett's neoplasia using volumetric laser endomicroscopy. Gastrointest Endosc. 2017 Nov;86(5):839-846. doi: 10.1016/j.gie.2017.03.011. Epub 2017 Mar 16. PMID 28322771
- [Background] Alvarez Herrero L, Curvers WL, van Vilsteren FG, Wolfsen H, Ragunath K, Wong Kee Song LM, Mallant-Hent RC, van Oijen A, Scholten P, Schoon EJ, Schenk EB, Weusten BL, Bergman JG. Validation of the Prague C&M classification of Barrett's esophagus in clinical practice. Endoscopy. 2013 Nov;45(11):876-82. doi: 10.1055/s-0033-1344952. Epub 2013 Oct 28. PMID 24165812
- [Background] The Paris endoscopic classification of superficial neoplastic lesions: esophagus, stomach, and colon: November 30 to December 1, 2002. Gastrointest Endosc. 2003 Dec;58(6 Suppl):S3-43. doi: 10.1016/s0016-5107(03)02159-x. No abstract available. PMID 14652541

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 133 of 148 subjects were randomized during their EGD procedure. Of those not randomized, 8 subjects had a segment of Barrett's esophagus less than 2cm, 3 subjects had esophagitis (LA Grade B or higher), and 4 subjects did not have a complete VLE exam due to technical malfunctions with the device.
Period: Overall Study
Arm/Group | VLE Without IRIS, Followed by VLE With IRIS | VLE With IRIS, Followed by VLE Without IRIS
Started | 67 | 66
Completed | 67 | 66
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VLE Without IRIS, Followed by VLE With IRIS | VLE With IRIS, Followed by VLE Without IRIS | Total
Number analyzed (Participants) | 67 | 66 | 133
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 28 | 60
  >=65 years | 35 | 38 | 73
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 18 | 42
  Male | 43 | 48 | 91
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time for Image Interpretation (Mean)
Description: The length of time required to fully assess and interpret the results of a VLE scan. Time will be a surrogate for ease of interpretation. Time will be recorded from start of image interpretation to the end of image interpretation. Length of the Barrett's segment will be taken into account (time per cm of Barrett's) when comparing this outcome between patients and procedures.
Time Frame: Index procedure, up to 1 hour
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | VLE Without IRIS, Followed by VLE With IRIS | VLE With IRIS, Followed by VLE Without IRIS
Number analyzed (Participants) | 67 | 66
Minutes
  Total interpretation time (VLE/IRIS) | 4.0 (3.75) | 4.6 (3.43)
  Interpretation time (VLE alone) | 3.8 (2.08) | 2.4 (2.10)
  First Interpretation Time | 3.8 (2.08) | 4.6 (3.43)
  Second Interpretation Time | 4.0 (3.75) | 2.4 (1.5)

2. Primary Outcome: Time for Image Interpretation (Mean - Scaled)
Description: as for outcome 1
Time Frame: Index procedure, up to 1 hour
Measure: Mean (Standard Deviation); unit: Centimeters/Minutes
Arm/Group | VLE Without IRIS, Followed by VLE With IRIS | VLE With IRIS, Followed by VLE Without IRIS
Number analyzed (Participants) | 67 | 66
Centimeters/Minutes
  Scaled First Interpretation Time | 1.2 (0.86) | 1.1 (0.62)
  Scaled Second Interpretation Time | 1.3 (1.25) | 0.6 (0.47)

3. Primary Outcome: Time for Image Interpretation (Median - Scaled)
Description: The length of time required to fully assess and interpret the results of a VLE scan. Time will be a surrogate for ease of interpretation. Time will be recorded from start of image interpretation to the end of image interpretation. Length of Barrett's will be taken into account (time per cm of Barrett's) when comparing this outcome between patients and procedures.
Time Frame: Index procedure, up to 1 hour
Measure: Median (Standard Deviation); unit: Centimeters/Minutes
Arm/Group | VLE Without IRIS, Followed by VLE With IRIS | VLE With IRIS, Followed by VLE Without IRIS
Number analyzed (Participants) | 67 | 66
Centimeters/Minutes
  Scaled First Interpretation Time | 1.0 (0.86) | 1.0 (0.62)
  Scaled Second Interpretation Time | 1.0 (1.25) | 0.5 (0.47)

4. Secondary Outcome: Subjects With Dysplasia on Biopsies
Description: Biopsy yield (in terms of dysplasia present versus not present) of subjects with IRIS biopsies (double laser mark) will be compared to subjects with VLE without IRIS biopsies (single laser mark) and subjects with random biopsies (taken every 1cm in a four quadrant fashion throughout the length of the Barrett's).
Time Frame: Index procedure
Measure: Number; unit: Participants with dysplasia on biopsies
Groups:
- VLE Without IRIS: VLE (Volumetric laser endomicroscopy) performed alone,
  VLE (Volumetric laser endomicroscopy): VLE uses infrared light to produce real time high-resolution cross sectional imaging of the esophagus.
- VLE With IRIS: VLE (Volumetric laser endomicroscopy) performed with IRIS (Intelligent real-time image segmentation) imaging.
  VLE (Volumetric laser endomicroscopy): VLE uses infrared light to produce real time high-resolution cross sectional imaging of the esophagus.
  IRIS (Intelligent real-time image segmentation): IRIS has the ability to identify and display three specific images features that may correlate with dysplasia that are represented in different color schemes.
- Seattle Protocol: Standardized method of biopsy collection entailing taking biopsies every 1cm of the Barrett's segment in a 4 quadrant fashion, the current standard of care.
Arm/Group | VLE Without IRIS | VLE With IRIS | Seattle Protocol
Number analyzed (Participants) | 133 | 133 | 100
Participants with dysplasia on biopsies | 29 | 34 | 24

ADVERSE EVENTS:
Time Frame: 1 week
Groups:
- VLE Without IRIS: VLE (Volumetric laser endomicroscopy) performed alone, followed by IRIS (Intelligent real-time image segmentation) imaging.
  IRIS (Intelligent real-time image segmentation): IRIS has the ability to identify and display three specific images features that may correlate with dysplasia that are represented in different color schemes.
  VLE (Volumetric laser endomicroscopy): VLE uses infrared light to produce real time high-resolution cross sectional imaging of the esophagus.
- VLE With IRIS: VLE (Volumetric laser endomicroscopy) performed with IRIS (Intelligent real-time image segmentation) imaging, followed by VLE alone.
  IRIS (Intelligent real-time image segmentation): IRIS has the ability to identify and display three specific images features that may correlate with dysplasia that are represented in different color schemes.
  VLE (Volumetric laser endomicroscopy): VLE uses infrared light to produce real time high-resolution cross sectional imaging of the esophagus.
Arm/Group | VLE Without IRIS | VLE With IRIS
All-Cause Mortality (participants affected / at risk) | 0/133 | 0/133
Serious Adverse Events (participants affected / at risk) | 0/133 | 0/133
Other Adverse Events (participants affected / at risk) | 0/133 | 0/133

LIMITATIONS AND CAVEATS:
By utilizing expert users, we're unable to assess the impact of IRIS on novice interpretation. We also utilized a surveillance biopsy protocol that avoided areas of laser marking to avoid confounding and were thus unable to compare VLE-related dysplasia detection to that which would have occurred in the standardized biopsy protocol. Finally, although we did randomize the order of interpretation, it is not possible to eliminate all bias from a subjective interpretation paradigm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT03814824/Prot_SAP_000.pdf